CLINICAL TRIAL: NCT00729183
Title: A Phase III Randomized, Placebo-Controlled Study to Evaluate the Effect of Odanacatib (MK-0822) on Bone Mineral Density (BMD) and Overall Safety, and to Estimate the Effect of Odanacatib (MK-0822) on Bone Micro-architecture in Postmenopausal Women Treated With Vitamin D
Brief Title: Study to Evaluate Efficacy of Odanacatib (MK-0822) on Bone Mineral Density (BMD) and Bone Micro-architecture and Overall Safety in Postmenopausal Women (MK-0822-031)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-031; 2008_539 (Other: Merck Registration Number)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib; Cholecalciferol; Calcium Carbonate; Calcium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Odanacatib 50 mg (Experimental): Participants receive 50 mg odanacatib and open-label 5600 IU vitamin D3 tablets once weekly for 24 months. Participants also receive 500 mg of open-label daily calcium supplement as needed to ensure a total daily calcium intake of 1200 mg.
  Interventions: Drug: Odanacatib; Drug: Vitamin D3; Drug: Calcium supplement
- Placebo (Placebo Comparator): Participants receive matching placebo to odanacatib and open-label 5600 IU vitamin D3 once weekly for 24 months. Participants also receive 500 mg of open-label daily calcium supplement as needed to ensure a total daily calcium intake of 1200 mg.
  Interventions: Drug: Placebo; Drug: Vitamin D3; Drug: Calcium supplement

INTERVENTIONS:
Drug: Odanacatib — Odanacatib 50 mg tablets, taken orally once weekly for 24 months.
  Other Names: MK-0822
  Arms: Odanacatib 50 mg
Drug: Placebo — Matching placebo tablets to odanacatib taken orally once weekly for 24 months.
  Arms: Placebo
Drug: Vitamin D3 — Vitamin D3 tablets (5600 IU) taken orally once weekly for 24 months.
Drug: Calcium supplement — Calcium supplement 500 mg tablet taken orally once daily (up to ~1200 mg total) for 24 months.
  Other Names: calcium carbonate; calcium citrate

SUMMARY:
This study will evaluate the safety and treatment effect of 50 mg odanacatib (MK-0822) with Vitamin D versus placebo with Vitamin D in postmenopausal women with low bone density. The primary efficacy hypothesis is that odanacatib will increase aBMD at the lumbar spine compared to placebo at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been postmenopausal for 3 years
* Participant has BMD t-score at the total hip, hip trochanter, femoral neck, or lumbar spine ≥ -1.5 but > -3.5
* Participant has 2 hips that are evaluable by dual-energy X-ray absorptiometry (DXA) and quantitative computed tomography (QCT), e.g. contain no hardware from orthopedic procedures
* Participant is ambulatory

Exclusion Criteria:

* Participant has had a previous hip fracture
* Participant has had >1 prior clinical vertebral fracture AND is a candidate for osteoporosis therapy
* Participant has been treated with oral bisphosphonates, strontium, parathyroid hormone (PTH) or other agents with an effect on bone
* Participant has had metabolic bone disorder other than osteoporosis
* Participant has renal stones, Parkinson's disease, multiple sclerosis (MS) or active parathyroid disease.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2010-03-23 (Actual); Study Completion 2011-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Engelke K, Fuerst T, Dardzinski B, Kornak J, Ather S, Genant HK, de Papp A. Odanacatib treatment affects trabecular and cortical bone in the femur of postmenopausal women: results of a two-year placebo-controlled trial. J Bone Miner Res. 2015 Jan;30(1):30-8. doi: 10.1002/jbmr.2292. PMID 24898537
- [Derived] Brixen K, Chapurlat R, Cheung AM, Keaveny TM, Fuerst T, Engelke K, Recker R, Dardzinski B, Verbruggen N, Ather S, Rosenberg E, de Papp AE. Bone density, turnover, and estimated strength in postmenopausal women treated with odanacatib: a randomized trial. J Clin Endocrinol Metab. 2013 Feb;98(2):571-80. doi: 10.1210/jc.2012-2972. Epub 2013 Jan 21. PMID 23337728

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 214 participants who met inclusion criteria were randomized into either the Odanacatib 50 mg arm (N=109) or the Placebo arm (N=105).
Groups:
- Odanacatib 50 mg: Participants received 50 mg odanacatib and open-label 5600 IU vitamin D3 tablets once weekly for 24 months. Participants also received 500 mg of open-label daily calcium supplement as needed to ensure a total daily calcium intake of 1200 mg.
- Placebo: Participants received matching placebo to odanacatib and open-label 5600 IU vitamin D3 once weekly for 24 months. Participants also received 500 mg of open-label daily calcium supplement as needed to ensure a total daily calcium intake of 1200 mg.
Period: Overall Study
Arm/Group | Odanacatib 50 mg | Placebo
Started | 109 | 105
Completed | 84 (Completed 24 month visit) | 90 (Completed 24 month visit)
Not Completed | 25 | 15
Not completed — Adverse Event | 11 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Odanacatib 50 mg | Placebo | Total
Number analyzed (Participants) | 109 | 105 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.3) | 64.0 (6.2) | 64.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 105 | 214
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 12 in Lumbar Spine Areal Bone Mineral Density (aBMD)
Description: aBMD (g/cm^2) was measured by dual-energy X-ray absorptiometry (DXA) at the lumbar spine and mean BMD measurements from at least 3 evaluable lumbar spine vertebrae (L1-L4) were used. If a vertebra was fractured at baseline or became fractured during the study, its BMD measurement was excluded from the analysis and the lumbar spine BMD was recalculated based on the three remaining vertebrae. aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the lumbar spine was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal Analysis of Covariates (ANCOVA) model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as primary and secondary outcome measures, respectively.
Time Frame: Baseline, 12 months
Population: Full-Analysis-Set (FAS) population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having Month 12 post-randomization lumbar spine aBMD endpoint data subsequent to at least one dose of study treatment, and having lumbar spine aBMD baseline (BL) data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 97
percent change | 3.63 [3.04 to 4.21] | 0.14 [-0.45 to 0.72]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; A longitudinal ANCOVA was used to obtain an estimate of the between-treatment difference in aBMD together with its 95% confidence interval (CI). The model, applied on all time points during treatment (Screening Visit [BL], Month 6, Month 12, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and BL value as covariate. The weighted Least Squares (LS) mean is based on the described model. Difference in LS Means = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis (LDA) Model; Difference in LS Means = 3.49, 95% CI 2-sided [2.66 to 4.32]

2. Primary Outcome: Percentage of Participants That Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's products, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The percentage of participants that experienced at least one AE was reported for each treatment arm.
Time Frame: Up to ~14 days post study end (up to ~24 months)
Population: All-Participants-as-Treated (APaT) population: all participants who took at least one dose of study medication, counted in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 109 | 105
percentage of participants | 82.6 | 84.8
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Estimated difference (versus Placebo) and CI were based on the Miettinen & Nurminen method; Test type: Superiority or Other; Difference in Percentage = -2.2, 95% CI 2-sided [-12.3 to 7.9]

3. Primary Outcome: Percentage of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's products, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The percentage of participants that discontinued study treatment (different from discontinuation of the study) due to an AE was reported for each treatment arm.
Time Frame: Up to ~14 days post study end (up to ~24 months)
Population: APaT population: all participants who took at least one dose of study medication, counted in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 109 | 105
percentage of participants | 10.1 | 5.7
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Estimated difference (versus Placebo) and CI were based on the Miettinen & Nurminen method; Test type: Superiority or Other; Difference in Percentage = 4.4, 95% CI 2-sided [-3.2 to 12.3]

4. Secondary Outcome: Percent Change From Baseline to Month 24 in Lumbar Spine aBMD
Description: aBMD (g/cm^2) was measured by DXA at the lumbar spine and mean BMD measurements from at least 3 evaluable vertebrae from L1 through L4 were used. If a vertebra was fractured at baseline or became fractured during the study, its BMD measurement was excluded from the analysis and the lumbar spine BMD was recalculated based on the three remaining vertebrae. aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the lumbar spine was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as primary and secondary outcome measures, respectively.
Time Frame: Baseline, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having Month 24 post-randomization lumbar spine aBMD endpoint data subsequent to at least one dose of study treatment, and having lumbar spine aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 90
percent change | 5.02 [4.28 to 5.76] | -0.38 [-1.09 to 0.34]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; A longitudinal ANCOVA model was used to obtain an estimate of the between-treatment difference in aBMD together with its 95% CI. The model, applied on all time points during treatment (Screening Visit [Baseline], Month 6, Month 12, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and BL value as covariate. The weighted LS mean is based on the described model. Difference in LS Means = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 5.39, 95% CI 2-sided [4.36 to 6.42]

5. Secondary Outcome: Percent Change From Baseline in Total Hip aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the total hip. All measurements utilized the same hip and at least 2 vertebrae for all time points. The left hip only was scanned. If the left hip was unevaluable, then the right hip was scanned. Once the appropriate leg was identified for scanning, it was used for all subsequent measurements. aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the total hip was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization total hip aBMD endpoint data subsequent to at least one dose of study treatment, and having total hip aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 97
percent change
  Month 12 (n=96, n=97) | 1.41 [0.92 to 1.89] | -0.16 [-0.64 to 0.32]
  Month 24 (n=82, n=90) | 2.43 [1.76 to 3.10] | -0.89 [-1.55 to -0.24]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; MONTH 12: A longitudinal ANCOVA model was used to obtain an estimate of the between-treatment difference in aBMD together with its 95% CI. The model, applied on all time points during treatment (Screening Visit [Baseline], Month 6, Month 12, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and baseline value as covariate. The weighted LS mean is based on the described model. Difference in LS Means at Month 12 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 1.57, 95% CI 2-sided [0.88 to 2.25]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; MONTH 24: A longitudinal ANCOVA model was used to obtain an estimate of the between-treatment difference in aBMD together with its 95% CI. The model, applied on all time points during treatment (Screening Visit [Baseline], Month 6, Month 12, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and baseline value as covariate. The weighted LS mean is based on the described model. Difference in LS Means at Month 24 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 3.32, 95% CI 2-sided [2.39 to 4.26]

6. Secondary Outcome: Percent Change From Baseline in Femoral Neck aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the femoral neck (hip). All measurements utilized the same hip and at least 2 vertebrae for all time points. The left hip only was scanned. If the left hip was unevaluable, then the right hip was scanned. Once the appropriate leg was identified for scanning, it was used for all subsequent measurements. aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the femoral neck was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization femoral neck aBMD endpoint data subsequent to at least one dose of study treatment, and having femoral neck aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 97
percent change
  Month 12 (n=96, n=97) | 1.03 [0.41 to 1.65] | -0.45 [-1.07 to 0.17]
  Month 24 (n=82, n=90) | 2.47 [1.67 to 3.28] | -1.33 [-2.11 to -0.56]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.001, LDA; Difference in LS Means = 1.48, 95% CI 2-sided [0.60 to 2.35]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 3.81, 95% CI 2-sided [2.69 to 4.93]

7. Secondary Outcome: Percent Change From Baseline in Hip Trochanter aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the hip trochanter. All measurements utilized the same hip and at least 2 vertebrae for all time points. The left hip only was scanned. If the left hip was unevaluable, then the right hip was scanned. Once the appropriate leg was identified for scanning, it was used for all subsequent measurements. aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the hip trochanter was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization hip trochanter aBMD endpoint data subsequent to at least one dose of study treatment, and having hip trochanter aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 97
percent change
  Month 12 (n=96, n=97) | 2.37 [1.59 to 3.15] | 0.18 [-0.60 to 0.95]
  Month 24 (n=82, n=90) | 4.75 [3.75 to 5.76] | -0.73 [-1.71 to 0.25]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 2.19, 95% CI 2-sided [1.09 to 3.29]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 5.48, 95% CI 2-sided [4.08 to 6.89]

8. Secondary Outcome: Percent Change From Baseline in Total Radius aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the total radius (forearm). aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the total radius was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization total radius aBMD endpoint data subsequent to at least one dose of study treatment, and having total radius aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 96
percent change
  Month 12 (n=96, n=96) | 0.01 [-0.44 to 0.47] | -0.70 [-1.15 to -0.24]
  Month 24 (n=82, n=90) | -0.19 [-0.71 to 0.34] | -1.89 [-2.40 to -1.38]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.030, LDA; Difference in LS Means = 0.71, 95% CI 2-sided [0.07 to 1.35]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 1.70, 95% CI 2-sided [0.97 to 2.43]

9. Secondary Outcome: Percent Change From Baseline in Ultradistal Radius aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the ultradistal radius (forearm). aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the ultradistal radius was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization ultradistal radius aBMD endpoint data subsequent to at least one dose of study treatment, and having ultradistal radius aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 96
percent change
  Month 12 (n=96, n=96) | 0.98 [0.25 to 1.70] | -0.73 [-1.46 to -0.01]
  Month 24 (n=82, n=90) | 1.25 [0.48 to 2.03] | -1.45 [-2.20 to -0.69]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.001, LDA; Difference in LS Means = 1.71, 95% CI 2-sided [0.69 to 2.73]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 2.70, 95% CI 2-sided [1.62 to 3.78]

10. Secondary Outcome: Percent Change From Baseline in Distal Radius aBMD
Description: aBMD (g/cm^2) data was measured by DXA at the one-third distal radius (forearm). aBMD data was centrally evaluated and all areal BMD measurements included a longitudinal BMD correction factor as determined by the quality control center. aBMD at the distal radius was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization distal radius aBMD endpoint data subsequent to at least one dose of study treatment, and having distal radius aBMD baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 96 | 96
percent change
  Month 12 (n=96, n=96) | -0.21 [-0.77 to 0.35] | -0.37 [-0.92 to 0.19]
  Month 24 (n=82, n=90) | -0.57 [-1.25 to 0.12] | -1.79 [-2.46 to -1.12]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.697, LDA; Difference in LS Means = 0.16, 95% CI 2-sided [-0.63 to 0.95]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.013, LDA; Difference in LS Means = 1.22, 95% CI 2-sided [0.27 to 2.18]

11. Secondary Outcome: Percent Change From Baseline in Trabecular Volumetric Bone Mineral Density (vBMD) at Central Section of Spine (L1)
Description: Trabecular vBMD at the lumbar spine (L1) was measured by quantitative computed tomography (QCT). All QCT-derived vBMD measurements were evaluated centrally (and possibly locally) for bone and soft tissue abnormalities. Trabecular vBMD at the lumbar spine (L1) was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization QCT spine (L1) endpoint data subsequent to at least one dose of study treatment, and having QCT spine (L1) baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 82 | 86
percent change
  Month 12 (n=82, n=86) | 6.58 [5.17 to 7.99] | -1.43 [-2.81 to -0.04]
  Month 24 (n=72, n=79) | 6.44 [4.64 to 8.24] | -5.02 [-6.76 to -3.28]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 8.01, 95% CI 2-sided [6.03 to 9.99]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 11.46, 95% CI 2-sided [8.96 to 13.97]

12. Secondary Outcome: Percent Change From Baseline in Trabecular vBMD at Central Section of Spine (L2)
Description: Trabecular vBMD at the lumbar spine (L2) was measured by quantitative computed tomography (QCT). All QCT-derived vBMD measurements were evaluated centrally (and possibly locally) for bone and soft tissue abnormalities. Trabecular vBMD at the lumbar spine (L2) was assessed at the Screening visit (Baseline), Month 6, Month 12, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures.
Time Frame: Baseline, 12 months, 24 months
Population: FAS population: a subset of All Randomized Participants with participants receiving at least one dose of study treatment, having post-randomization QCT spine (L2) endpoint data subsequent to at least one dose of study treatment, and having QCT spine (L2) baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 84 | 86
percent change
  Month 12 (n=84, n=86) | 5.67 [4.32 to 7.02] | -0.00 [-1.34 to 1.34]
  Month 24 (n=73, n=79) | 5.97 [4.25 to 7.68] | -3.41 [-5.08 to -1.74]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 5.68, 95% CI 2-sided [3.77 to 7.58]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = 9.38, 95% CI 2-sided [6.98 to 11.77]

13. Secondary Outcome: Percent Change From Baseline in Serum C-Terminal Telopeptides of Type 1 Collagen (s-CTx) Level
Description: s-CTx is a biochemical marker index of bone resorption. s-CTx was measured via fasting blood draws at Baseline (Randomization), Month 6, Month 12, Month 18, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures. S-CTx was analyzed using the log-transformed fraction from baseline using the per-protocol approach. Data were back-transformed for presentation and geometric LS mean percent change from baseline was reported with 95% CI.
Time Frame: Baseline, 12 months, 24 months
Population: Per-Protocol (PP) population: All participants receiving at least one dose of study treatment and with available s-CTx data, excluding participants with important deviations from the protocol that may have substantially affected the results.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 89 | 87
percent change
  Month 12 (n=89, n=87) | -53.33 [-57.62 to -48.61] | 0.70 [-8.70 to 11.07]
  Month 24 (n=74, n=78) | -42.56 [-50.27 to -33.65] | 3.03 [-10.57 to 18.69]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; MONTH 12: A longitudinal ANCOVA model was used to obtain geometric LS mean percent change from BL in s-CTx (back-transformation of the log-transformed fraction from BL) and its 95% CI. The model, applied on all time points during treatment (Baseline [Randomization], Month 6, Month 12, Month 18, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and baseline value as covariate. Difference in LS Means at Month 12 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = -54.03, 95% CI 2-sided [-64.81 to -43.26]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; MONTH 24: A longitudinal ANCOVA model was used to obtain geometric LS mean percent change from BL in s-CTx (back-transformation of the log-transformed fraction from BL) and its 95% CI. The model, applied on all time points during treatment (Baseline [Randomization], Month 6, Month 12, Month 18, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and baseline value as covariate. Difference in LS Means at Month 12 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = -45.59, 95% CI 2-sided [-62.22 to -28.96]

14. Secondary Outcome: Percent Change From Baseline in Serum N-Terminal Propeptides of Type 1 Collagen (s-P1NP) Level
Description: s-P1NP is a biochemical marker index of bone formation. s-P1NP was measured via fasting blood draws at Baseline (Randomization), Month 6, Month 12, Month 18, and Month 24 for the repeated measures longitudinal ANCOVA model, with percent change from baseline at Months 12 and 24 pre-specified to be reported as secondary outcome measures. s-P1NP was analyzed using the log-transformed fraction from baseline using the per-protocol approach. Data were back-transformed for presentation and geometric LS mean percent change from baseline was reported with 95% CI.
Time Frame: Baseline, 12 months, 24 months
Population: PP population: All participants receiving at least one dose of study treatment and with available s-P1NP data, excluding participants with important deviations from the protocol that may have substantially affected the results.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 90 | 88
percent change
  Month 12 (n=90, n=88) | -28.32 [-35.30 to -20.58] | -2.97 [-12.57 to 7.69]
  Month 24 (n=76, n=80) | -11.06 [-20.40 to -0.61] | -1.99 [-12.32 to 9.56]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; MONTH 12: A longitudinal ANCOVA model was used to obtain geometric LS mean percent change from BL in s-P1NP (back-transformation of the log-transformed fraction from BL) and its 95% CI. The model, applied on all time points during treatment (Baseline [Randomization], Month 6, Month 12, Month 18, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and BL value as covariate. Difference in LS Means at Month 12 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p < 0.001, LDA; Difference in LS Means = -25.34, 95% CI 2-sided [-37.77 to -12.92]
Statistical Analysis 2: Comparison: Odanacatib 50 mg vs Placebo; MONTH 24: A longitudinal ANCOVA model was used to obtain geometric LS mean percent change from BL in s-P1NP (back-transformation of the log-transformed fraction from BL) and its 95% CI. The model, applied on all time points during treatment (Baseline [Randomization], Month 6, Month 12, Month 18, Month 24), included treatment, region, time and interaction between treatment and time as fixed effects, and BL value as covariate. Difference in LS Means at Month 24 = Odancatib 50 mg minus Placebo; Test type: Superiority or Other; p = 0.225, LDA; Difference in LS Means = -9.07, 95% CI 2-sided [-23.69 to 5.56]

ADVERSE EVENTS:
Time Frame: ~14 days post study end (up to ~24 months)
Description: APaT population: all participants who took at least one dose of study medication, counted in the treatment group corresponding to the study treatment they actually received.
Arm/Group | Odanacatib 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 13/109 | 16/105
Other Adverse Events (participants affected / at risk) | 67/109 | 68/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg (N=109) | Placebo (N=105)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg (N=109) | Placebo (N=105)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (6)
Bronchitis (Infections and infestations) | 2 (2) | 7 (9)
Cystitis (Infections and infestations) | 5 (6) | 6 (9)
Influenza (Infections and infestations) | 10 (10) | 6 (6)
Nasopharyngitis (Infections and infestations) | 15 (18) | 8 (10)
Urinary tract infection (Infections and infestations) | 8 (11) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (19) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 16 (19)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9) | 8 (10)
Headache (Nervous system disorders) | 6 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 9 (12)
Hypertension (Vascular disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.